CLINICAL TRIAL: NCT06650397
Title: Absorption of Zinc and Iron from Nixtamalized Biofortified Maize in School-aged Children in Guatemala
Brief Title: Guatemala Biofortified Maize Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Institute of Nutrition of Central America and Panama (Other); Semilla Nueva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24-1030; 7200AA23FA00027 (Other Grant/Funding Number: U.S. Agency for International Development)
Record Dates: First submitted 2024-09-04; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Zinc Absorption; Iron Absorption
Keywords: biofortification; stable isotope; maize; Guatemala; school-aged children
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biofortified maize (Experimental): Children consume biofortified maize that has been traditionally bred to have higher amounts of iron and zinc. Children consume the biofortified maize via 10-15 tortillas a day for 3 days.
  Interventions: Other: Biofortified maize
- Traditional Maize (Placebo Comparator): Children consume traditional maize that has lower amounts of iron and zinc compared to the biofortified maize. Children consume the maize via 10-15 tortillas a day for 3 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Biofortified maize — Maize that has been grown to have higher amounts of iron and zinc.
  Arms: Biofortified maize
Other: Placebo — Traditional maize
  Arms: Traditional Maize

SUMMARY:
Zinc (Zn) and iron (Fe) deficiencies are common in Guatemala, and maize is a staple food throughout the country. The primary aim of this study is to demonstrate if utilizing nixtamalized biofortified maize has the potential to increase dietary Zn and Fe intake and improve the amount of Zn and Fe absorbed when compared to diets incorporating traditional maize (control). This is a randomized, double blinded, comparison study of biofortified vs control maize prepared as tortillas from nixtamalized masa. This study will enroll up to 56 school aged children (10-14 yrs old) living in agricultural communities in the Western Highlands of Guatemala (28/group x 2 groups). Researchers will utilize Zn and Fe stable isotopes to measure total absorbed Zn and Fe. Participants will be active in the study for 27 days. During this time, they will have anthropometric measurements taken and collect 2 blood samples, 1 stool sample, and 9 urine samples.

ELIGIBILITY:
Inclusion criteria:

* 10-14 years old school children (male and female sex)
* BMI between10-85%tile
* Typically eat homemade tortillas at each meal every day

Exclusion criteria:

* Taking iron or zinc supplements
* Hemoglobin less than 12.9 g/dl for children 10-11 yrs old and less than13.4 g/dl for children 12-14 yrs old (Per the WHO's 2024 publication hemoglobin cut-offs for identifying anemia are 5-11 yrs: less than 11.5 g/dl; 12-14 yrs: less than 12.0 g/dl. To adjust for the elevation of Tecpán at 2254 m, 1.4 g/dl is added to the cut-off point.)
* Girls who are having a menstrual period during the metabolic studies

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Total absorbed iron (TAI) (mg) | 2 days
  Total absorbed iron from the diet = fractional absorption of iron x total dietary iron (mg)
Total absorbed zinc (TAZ) (mg) | 1 day
  Total zinc absorbed from the diet = fractional absorption of zinc x total dietary zinc (mg)

SECONDARY OUTCOMES:
Plasma C-reactive protein (CRP) (mg/dL) | 1 day
  CRP is used to measure systemic inflammation
Plasma zinc concentration (mcg/dL) | 1 day
  Plasma zinc concentration is used to assess zinc status
Plasma Alpha(1)-acid glycoprotein (AGP) (mg/dL) | 1 day
  AGP is used to measure systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Institute of Nutrition of Central America and Panama, Guatemala City, Departamento de Guatemala, Guatemala

IPD SHARING:
Plan to Share IPD: Undecided
A de-identified dataset will be made available upon request.